CLINICAL TRIAL: NCT00501553
Title: Vitamin D in Patients With Heart Failure
Acronym: KarViD
Status: Completed | Type: Observational
Sponsor: Hvidovre University Hospital (Other)
Other Study IDs: 2005-41-5263; (KF)01 264904
Record Dates: First submitted 2007-07-13; First posted 2007-07-16 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2007-07

CONDITIONS: Heart Failure
Keywords: Heart Failure,; Vitamin D status,; NT-proBNP
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
To investigate the prevalence of vitamin D deficiency in patients with Heart Failure.

To investigate if vitamin D levels are correlated to the degree of Heart Failure.

ELIGIBILITY:
Inclusion Criteria:

* Patient in the Heart Failure Clinic, Hvidovre Hospital
* Willing to participate and sign informed consent over 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Heart Failure patients
Sampling Method: Probability Sample
Enrollment: 148 (Actual)
Dates: Start 2005-06; Study Completion 2007-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Louise L Schierbeck, MD, Principal Investigator — Hvidovre UH; Jens-Erik B Jensen, MD, PhD, Study Chair — Hvidovre UH
Locations (1):
- Hvidovre University Hospital, Hvidovre, Denmark